CLINICAL TRIAL: NCT03799952
Title: A Randomized Control Trial - Zoomers for the Capital Region: A Peer-Led Exercise Program for Aging Adults
Brief Title: Zoomers for the Capital Region: A Peer-Led Exercise Program for Aging Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of New Brunswick (Other)
Collaborators: New Brunswick Health Research Foundation (Other); Horizon Health Network (Other); Universite de Moncton (Other); Fitness New Brunswick (Other)
Responsible Party: Principal Investigator, Danielle Bouchard, Associate Professor, University of New Brunswick
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2019-01Zoom
Record Dates: First submitted 2018-12-20; First posted 2019-01-10 (Actual); Results first posted 2021-07-14 (Actual); Last update posted 2021-07-14 (Actual); Status verified 2021-07

CONDITIONS: Aging; Fall
Keywords: Older adult; Peer-led exercise program; Risk of falling

STUDY DESIGN:
Intervention Model Description: Randomized to a control or intervention group. The intervention group will have pre- and post-testing following 12-weeks of exercise, while the control group will have pre- and post-testing following 12-weeks of "normal" activity.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Participants are offered to attend a 12-week exercise program, classes offered twice a week, each class 60 minutes in length.
  Interventions: Behavioral: Zoomers on the Go Exercise Program
- Control (No Intervention): Participants are instructed to continue with their daily activities and their "normal" physical activity levels for 12-weeks.

INTERVENTIONS:
Behavioral: Zoomers on the Go Exercise Program — 60 minute exercise class involving resistance and aerobic training activities, as well as flexibility and balance activities. An educational handout is offered at the end of every class, relating to health behaviour.
  Arms: Intervention

SUMMARY:
The objective of this study is to recruit a group of older adults and study a broad set of physical health, mental health, and social outcomes when participants exercise with an older adult, peer-led exercise program.

The program to be evaluated is called Zoomers on the Go. It is a 12-week program which involves two 60-minute sessions per week and educates participants about falls, along with aerobic and resistance exercise, flexibility, and balance activities. The program is offered to older adults (age 50+) and it is delivered in their community by an older adult who is trained as a certified Zoomers group exercise leader.

Participants will be recruited, then randomized so that half of them can participate in a Zoomers class in the spring (intervention group) while half will have to wait until the fall of 2019 (control group). Pre-testing for both groups will begin around March 2019. The intervention group will participate in the program for 12 weeks, then there will be post-testing following this 12-weeks for both groups. Outcomes will be compared for the intervention and control groups, to determine if there are changes in the data pre- to post-measurements that are evident solely for the intervention group.

DETAILED DESCRIPTION:
This study is a randomized control trial where subjects will be randomly assigned to a control or an intervention group. Participants will be recruited through general advertisements (e.g. radio, newspaper, posters), in Fredericton and surrounding areas. These participants will be volunteers, and no compensation will be provided besides having access to a free exercise program in their community. Eligibility will be determined by the research staff prior to the baseline assessment day.Eligible participants will be evaluated at an initial day of testing at either a Horizon CommunityHealth Centre or at the University of New Brunswick in the Cardiometabolic Exercise and Lifestyle Laboratory (CELLab). This first visit will involve the confirmation of eligibility, reading and signing a consent form, and the administration of the measurements discussed previously. All research staff will have received the appropriate training to deliver these fitness assessments, finger pricks, and interviews.

At the end of the baseline visit, research staff will randomly assign participants to the intervention or control group. The participant will wear a pedometer for seven consecutive days following this initial visit. The paper form for any information collected (e.g. consent form) will be stored in the CELLab at UNB in a locked cabinet. The CELLab has limited access; only staff has access through a password to the lab. All information will be linked to a participant number for which the only linkable personal information (e.g., name, age, sex) will be kept in a password protected computer and only the Principal Investigator, Co-Investigators, and Research Coordinator will have access to this information. Information will be stored for a maximum of 7 years.

Following this baseline assessment, participants in the intervention group will be assigned to an exercise program most convenient to them. This is a 12-week exercise program, offered twice a week. Full attendance is not mandatory for being a participant. This is a peer-led exercise program, meaning it is instructed by a leader of similar age. This leader has received extensive Fitness New Brunswick training to deliver a program aimed to reduce the risk of falls and help older adults safely increase their physical activity levels. This 60-minute exercise program involves aerobic and resistance exercise, as well as flexibility and balance activities. The program is currently designed to help individuals meet the physical activity guidelines. Participants' numbers will be used to register attendance from the leaders.

Following this 12-week intervention or control period, participants will repeat all the baseline assessments (including questionnaires and interviews), with an exception that they will not have to wear the pedometer in the follow up visit. The primary objective will be to determine whether participants' experiences with the program were positive or negative, and specifically identifying participants' attributions of why/how the exercise intervention positively impacted their physical and/or mental health.

ELIGIBILITY:
Inclusion Criteria:

* 50 years of age or older
* Can exercise with minimal supervision (cleared for physical activity)
* Can commit to a 12-week exercise program (2 sessions/week)

Exclusion Criteria:

* Under 50 years of age
* Not cleared to perform physical activity

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2019-02-07 (Actual); Primary Completion 2019-11-28 (Actual); Study Completion 2019-11-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Kinesiology Building, Fredericton, New Brunswick, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bouchard DR, Olthuis JV, Bouffard-Levasseur V, Shannon C, McDonald T, Senechal M. Peer-led exercise program for ageing adults to improve physical functions - a randomized trial. Eur Rev Aging Phys Act. 2021 Feb 11;18(1):2. doi: 10.1186/s11556-021-00257-x. PMID 33573594

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment occurred between January and March 2019. Participants were recruited through radio advertisements, newspapers, posters, and social media. Per the participants availability they were allocated to the randomization or preferred arm.
Pre-assignment Details: Participants were excluded if they were not cleared by the Get Active Questionnaire and did not receive clearance from their primary physician to participate
Period: Overall Study
Arm/Group | Intervention | Control
Started | 31 | 31
Completed | 30 | 29
Not Completed | 1 | 2
Not completed — Program was too easy, discontinued | 1 | 0
Not completed — Lost to Follow-up | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention | Control | Total
Number analyzed (Participants) | 30 | 29 | 59
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.6 (7.2) | 66.1 (7.0) | 66.4 (7.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 23 | 51
  Male | 2 | 6 | 8
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Race/Ethnicity not collected Population: Not collected
Region of Enrollment [Number; unit: participants]
  Canada | 30 | 29 | 59
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 28.9 (4.5) | 25.8 (4.8) | 27.4 (4.9)
Occupation (Retired) [Count of Participants; unit: Participants] | 19 | 14 | 33
Marital Status (Married) [Count of Participants; unit: Participants] | 14 | 20 | 34
Household Income (>$100,000/year) [Count of Participants; unit: Participants] | 6.0 | 6.0 | 12
Physical Activity Level (Steps/day) [Mean (Standard Deviation); unit: Steps/day] | 6349 (2903) | 7221 (2964) | 6762 (2939)
Physical Activity Level (MVPA/week) [Mean (Standard Deviation); unit: Minutes of MVPA per week] | 68 (68) | 48 (81) | 58 (74)

OUTCOME MEASURES:

1. Primary Outcome: Balance
Description: One leg stand test (seconds)
Time Frame: Change pre and post (after the 12 weeks)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 30 | 29
score on a scale
  Pre (eyes open) | 26.7 (14.4) | 27.9 (16.4)
  Post (eyes open) | 34.7 (13.4) | 29.7 (15.6)
  Pre (eyes closed) | 5.0 (3.4) | 4.9 (3.2)
  Post (eyes closed) | 5.3 (3.5) | 4.4 (2.9)

2. Primary Outcome: Walking Speed
Description: 6-minute test (meters walked)
Time Frame: Change pre and post (after the 12 weeks)
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | Intervention | Control
Number analyzed (Participants) | 30 | 29
meters
  Pre | 476 (94.3) | 507 (90.3)
  Post | 539 (82.5) | 504 (79.7)

3. Primary Outcome: Flexibility
Description: Back scratch test (cm). The Back Scratch Test is a measure of flexibility of your upper body. Place your right hand behind your back with your palm out and your fingers extended up. Reach up as far as possible and attempt to touch the fingers of your two hands together. Some people are not able to touch at all, while others' fingers may overlap. Position fingers so that they are pointing toward each other. The distance between the fingertips of one hand and the other is measured to the nearest half-inch. If fingers overlap, the amount of the overlap will be measured. Fingertips just touching receive a score of "0". If fingers do not touch, it is a negative score of the distance between the fingers, measured to the nearest .5 or half inch. It is a positive score if fingers overlap, measuring the overlap to the nearest .5 or half inch.
Time Frame: Change pre and post (after the 12 weeks)
Measure: Mean (Standard Deviation); unit: centimeters
Arm/Group | Intervention | Control
Number analyzed (Participants) | 30 | 29
centimeters
  Pre | -7.5 (9.9) | -5.2 (9.7)
  Post | -5.7 (9.9) | -4.7 (9.9)

4. Primary Outcome: Strength, Arm Curl Test
Description: Number of bicep curls with light weight
Time Frame: Change pre and post (after the 12 weeks)
Measure: Mean (Standard Deviation); unit: reps/30 seconds
Arm/Group | Intervention | Control
Number analyzed (Participants) | 30 | 29
reps/30 seconds
  Pre | 20.1 (5.1) | 17.3 (4.1)
  Post | 23.9 (4.9) | 17.4 (3.5)

5. Primary Outcome: Strength, Chair Stand Test
Description: Chair stand test, number of chair stand in 30 seconds
Time Frame: Change pre and post (after the 12 weeks)
Measure: Mean (Standard Deviation); unit: reps/30 seconds
Arm/Group | Intervention | Control
Number analyzed (Participants) | 30 | 29
reps/30 seconds
  Pre | 14.1 (2.6) | 13.6 (2.7)
  Post | 17.9 (4.4) | 14.1 (3.5)

6. Secondary Outcome: Depression, Anxiety, Stress
Description: Depression Anxiety Stress Scales - 21 item (DASS-21) was used to measure past week depression, anxiety, and stress. Low is better. (Lovibond & Lovibond, 1995).
Time Frame: Pre and post (before and after the 12 week exercise program)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 30 | 29
score on a scale
  Pre Stress (0-28) | 6.0 (5.6) | 5.7 (6.2)
  Post Stress (0-28) | 4.1 (3.9) | 8.2 (7.7)
  Pre Anxiety (0-20) | 3.5 (3.8) | 2.6 (4.7)
  Post Anxiety (0-20) | 3.2 (3.3) | 5.0 (7.5)
  Pre Depression (0-34) | 4.8 (6.3) | 3.2 (3.8)
  Post Depression (0-34) | 3.2 (5.6) | 5.5 (9.1)

7. Secondary Outcome: Perceived Quality of Life
Description: The Short Form Health Survey - 36 items (SF-36) was used to measure day-to-day functioning and quality of life (Ware & Sherbourne, 1992). The scale is composed of eight domain subscales (i.e., Physical Functioning, Role Limitations due to Physical Health, Pain, General Health, Energy/Fatigue, Social Functioning, Role Limitations due to Emotional Problems, Emotional Well-Being) scored from 0 (worst) to 100 (excellent).
Time Frame: Pre and post (before and after the 12 week exercise program)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 30 | 29
score on a scale
  Pre Physical Functioning | 78.0 (21.2) | 80.9 (20.1)
  Post Physical Functioning | 81.2 (20.2) | 80.4 (18.8)
  Pre Limitations due to Physical Health | 78.3 (33.9) | 81.7 (28.8)
  Post Limitations due to Physical Health | 90.8 (24.1) | 79.0 (32.8)
  Pre Pain | 73.5 (22.3) | 79.1 (17.6)
  Post Pain | 71.9 (20.8) | 71.0 (23.0)
  Pre General Health | 71.2 (19.1) | 72.4 (11.8)
  Post General Health | 75.5 (15.6) | 69.8 (16.4)
  Pre Energy/Fatigue | 63.5 (19.1) | 67.4 (18.0)
  Post Energy/Fatigue | 68.7 (16.3) | 65.4 (17.6)
  Pre Social Functioning | 90.2 (14.9) | 88.9 (16.3)
  Post Social Functioning | 92.1 (13.7) | 86.4 (19.1)
  Pre Limitations Emotional Problems | 84.6 (28.3) | 78.8 (33.8)
  Post Limitations Emotional Problems | 88.9 (25.3) | 84.0 (32.1)
  Pre Emotional Well-Being | 80.4 (13.5) | 82.5 (12.4)
  Post Emotional Well-Being | 84.7 (10.2) | 78.7 (13.2)

8. Other Pre Specified Outcome: Researcher-generated Measure of Exercise Self-efficacy Based on Bandura's Concept of Self-efficacy
Description: The outcome measure on exercise self-efficacy (based on Bandura's concept of self-efficacy) is measured on a 1-4 scale. A higher score is more desirable than a lower score
Time Frame: Pre and post (before and after the 12 week exercise program)
Reporting Status: Not Posted

9. Other Pre Specified Outcome: Connectedness, Sense of Belonging, and Friendships
Description: All collected information via interviews with participants
Time Frame: Following the 12 week program
Reporting Status: Not Posted

10. Other Pre Specified Outcome: The Amount of Bodily Sway When Performing Tasks and Balancing.
Description: Measured by a portable biomechanical board. Can detect sway through sensors.
Time Frame: Pre and post (before and after the 12 week exercise program)
Reporting Status: Not Posted

11. Other Pre Specified Outcome: Blood Draw Via Finger Prick and Analyzed With a Cardiochek Machine
Description: Blood draw via finger prick and analyzed with a Cardiochek machine
  An individual's glucose levels in capillary blood, taken by a finger prick and assessed with a Cardiochek machine
Time Frame: Pre and post (before and after the 12 week exercise program)
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Intervention | Control
Number analyzed (Participants) | 30 | 29
mmol/L
  Pre | 5.34 (0.69) | 5.61 (1.05)
  Post | 4.70 (0.52) | 5.11 (0.65)

12. Other Pre Specified Outcome: Measured on a Portable Biomechanical Board.
Description: An individual's centre of mass as determined by sensors on a biomechanical board.
Time Frame: Pre and post (after the 12 weeks)
Reporting Status: Not Posted

13. Other Pre Specified Outcome: Systolic Blood Pressure
Description: Blood pressure cuff (mmHg)
Time Frame: Pre and post (after the 12 weeks)
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Intervention | Control
Number analyzed (Participants) | 30 | 29
mmHg
  Pre | 123.8 (12.6) | 127.5 (11.1)
  Post | 125.7 (14.9) | 124.5 (9.5)

14. Other Pre Specified Outcome: Resting Heart Rate
Description: Radial pulse palpation (bpm)
Time Frame: Pre and post (after the 12 weeks)
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | Intervention | Control
Number analyzed (Participants) | 30 | 29
beats per minute
  Pre | 68.1 (9.4) | 70.5 (6.7)
  Post | 63.0 (7.0) | 67.2 (7.6)

15. Other Pre Specified Outcome: Blood Draw Via Finger Prick and Analyzed With a Cardiochek Machine for Cholesterol Levels
Description: An individual's cholesterol levels in capillary blood, taken by a finger prick and assessed with a Cardiochek machine
Time Frame: Pre and post (before and after the 12 week exercise program)
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Adverse events were monitored from the beginning of the study, through to study completion.
Description: There were no adverse events that took place from the beginning to the end of the study.
Arm/Group | Intervention | Control
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/29
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/29
Other Adverse Events (participants affected / at risk) | 0/30 | 0/29

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-11-23): https://cdn.clinicaltrials.gov/large-docs/52/NCT03799952/Prot_SAP_000.pdf